CLINICAL TRIAL: NCT05801497
Title: Balneotherapy in Primary Fibromyalgia: Impact on Algo-functional Indexes, Quality of Life, and Anxio-depressive Symptoms
Brief Title: Balneotherapy in Primary Fibromyalgia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Siena (Other)
Collaborators: Azienda Ospedaliera Universitaria Senese (Other)
Responsible Party: Principal Investigator, fioravanti antonella, Scientific Coordinator, Azienda Ospedaliera Universitaria Senese
Other Study IDs: FIBROTHERM
Record Dates: First submitted 2023-03-22; First posted 2023-04-06 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Fibromyalgia, Primary
Keywords: balneotherapy
MeSH Terms: conditions — Fibromyalgia | interventions — Balneology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Balneotherapy Group: Patients will receive a cycle of BT or a cycle of mud-bath therapy once daily for 12 days for a total duration of two weeks, in addition to their usual treatments for fibromyalgia. The bath can be performed both in a bathube or in a pool for 10 minutes, at a 37-38°C. The application of mud will follow the standard procedure with a duration of 15-20 minutes at 40-45°C. After the treatment, patients will relax for 20-30°C minutes. To be included in the study, thermal interventions must be carried out with sulfourous, solfate, bicarbonate, saline or sodium chloride and arsenical-ferruginous mineral waters, according to the classification by Marotta and Sica.
  Interventions: Procedure: Balneotherapy
- Control Group: This group will include patients who will refuse the thermal treatment for personal reasons. Patients will continue their established routinary care for FS. The treatment must be stable for at least 3 months; some variations in analgesic consumption will be possible and will be collected in the clinical chart.

INTERVENTIONS:
Procedure: Balneotherapy — The patients in the BT group will be treated with 12 daily immersion in a bathtub or in a pool at a 37-38°C or with a combination of bath and mud-packs to carry out in a period of two weeks.
  The application of mud-packs will follow the standard procedure with a duration of 15-20 minutes at 40-45°C. After the treatment, patients will have 20-30 minutes of bed rest. To be included in the study, thermal interventions must be carried out with sulfourous, solfate, bicarbonate, saline or sodium chloride and arsenical-ferruginous mineral waters, according to the classification by Marotta and Sica.
  Groups: Balneotherapy Group

SUMMARY:
Balneotherapy (BT) is recommended as non-pharmacological treatment for Fibromyalgia Syndrome (FS). BT efficacy is based on beneficial properties of both mud bath and stay in a spa environment. The main aim of this multicentric prospective longitudinal cohort study is to evaluate BT effectiveness in patients withFS. All FS patients with a stable treatment in the past month and a Fibromyalgia Impact Questionnaire (FIQ) score ≥39 will be enrolled after providing written informed consent. Patients will be divided into two groups based on whether or not BT is added to usual therapy: BT Group and Control Group. Each patients will be assessed at baseline, after 15 and 45 days in BT Group and at baseline and after 15 days in Control group with an assessment of pain by Visual Analogue Scale, FIQ, Short-Form Health Survey, State-Trait Anxiety Inventory (STAI) and Center for Epidemiologic Studies Depression Scale (CES-D). Collected data will provide a new insight of BT role and the removal of daily stress in FS management

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary FS according to the 2010 American College of Rheumatology (ACR) criteria;
* Pharmacological and non pharmacological treatment stable for at least 3 months;
* FIQ-Total score ≥ 39

Exclusion Criteria:

* Secondary FS;
* Primary FS patients actually enrolled in other clinical trials;
* Patients who had receveid a cycle of BT or of mud-bath in the previous 6 months;
* Patients treated with intra-articular steroid injections of any joints in the previous 3 months;
* Pregnancy or breastfeeding;
* Cognitive or psychiatric disorders and history of substance abuse;
* Absolute and relative contraindications to BT

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants are stratified into two groups (BT Group and Control Group) based on whether or not balneotherapy or a cycle of bath combined with mud-packs will be added to the usual therapy for FS
Sampling Method: Probability Sample
Enrollment: 520 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Minimal Clinically Important Difference (MCID) | 15 days
  Percentage of patients achieving MCDI, defined as a reduction>14% of FIQ-total score

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) | basal time;15 days;45 days
  Assessment of pain on a 0-10-cm Visual Analogue Scale (VAS) with 0 = "no pain" and 10 = "the worst pain possible"
Fibromyalgia Impact Questionnaire (FIQ) | basal time;15 days;45 days
  FIQ is an extensively validated patient self-report questionnaire, evaluating the impact of FS on daily life. In this study, we will use the Italian version of the FIQ. It ranges from 0 to 100, with higher scores indicating greater impact of FS on functioning.
Short-Form Health Survey (SF-12) | basal time;15 days;45 days
  The 12-item SF-12 is a short version of SF-36 that is a widely used measure of health and well-being, validated in multiple countries, including Italy. SF-12 comprises two main domains: the physical component score (PCS) and the mental component score (MCS), and eight scales for assessing eight dimensions: physical functioning, physical role, social role, emotional role, bodily pain, general health, vitality, and mental health. Scores range from "0 to 100" where "0" indicates the worst condition and "100" indicates the best possible condition.
State-Trait Anxiety Inventory (STAI) | basal time;15 days;45 days
  STAI is a self-report questionnaire with two independent 20-item scales (STAI T-Anxiety Scale or Form X-2 and STAI S-Anxiety Scale or Form X-1) for measuring state-related or trait-related anxiety. A high score on the STAI corresponds to a high level of anxiety symptoms. We will use the Italian validated version.
Center for Epidemiologic Studies Depression Scale (CES-D) | basal time;15 days;45 days
  The 20-item CES-D Scale is frequently used to estimate the prevalence of depressive symptomatology in the general population. Respondents rate the frequency with which they have experienced particular depressive symptoms during the past week. Responses to each item range from 0 (less than 1 day) to 3 (5-7 days) and are summed to compute a total score. The Italian version measures one depression factor scoring from 0 to 60; scores of 16 or above are considered cases of depression.
Adverse events | 15 days
  Percentage of patients reporting adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera Universitaria Senese, Siena, Italy

IPD SHARING:
Plan to Share IPD: Undecided